CLINICAL TRIAL: NCT04305626
Title: Clinical Evaluation of the p64 MW HPC and the p48 MW HPC Flow Diverters in an Observational Registry
Brief Title: Coated Mongolian Aneurysm Treatment Study 1
Acronym: COMATS 1
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Phenox GmbH (Industry)
Responsible Party: Sponsor
Other Study IDs: STUD-192206
Record Dates: First submitted 2020-03-09; First posted 2020-03-12 (Actual); Last update posted 2022-04-26 (Actual); Status verified 2021-10

CONDITIONS: Intracranial Aneurysm; Aneurysm; Vascular Diseases
Keywords: p64 MW HPC; p48 MW HPC; Flow Diverter; HPC; Dual antiplatelet therapy; Outcome; Occlusion; Stroke
MeSH Terms: conditions — Intracranial Aneurysm; Aneurysm; Vascular Diseases; Bites and Stings; Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Endovascular treatment of intracranial aneurysms — Endovascular treatment of intracranial aneurysms with flow diversion.

SUMMARY:
The purpose of this study is to assess safety and effectiveness of the p64 MW HPC or p48 MW HPC Flow Modulation Device under Dual Antiplatelet Medication.

DETAILED DESCRIPTION:
Title: Observational Registry With p64 MW HPC and p48 MW HPC in Unruptured Anterior Circulation Aneurysms Under Dual Antiplatelet Medication.

Purpose: To assess safety and effectiveness of p64 MW HPC or p48 MW HPC under Dual Antiplatelet Medication in consecutive patients with unruptured anterior circulation aneurysms.

Follow-up intervals: Independent follow-ups (after 3 to 6 months and after 12 months and after 24 months) according to site specific standard.

ELIGIBILITY:
Inclusion Criteria:

* At least one unruptured sidewall aneurysm in the anterior circulation
* No implant (e.g., stent) in the target vessel segment
* Age >18 years and <80 years
* Not pregnant and in women of childbearing age, on oral contraception for two years following the procedure
* No participation in another trial
* No concomitant disease limiting the life expectancy to <2 years
* No allergy to non-ionic contrast medium or to ASA and P2Y12 receptor antagonists
* No other neurovascular disorder in the same vascular territory requiring treatment in the foreseeable future
* Ability and willingness to comply with the medication requirements within the study,
* Ability to understand the goal and risks of this study.

Exclusion Criteria:

* Intracranial aneurysm considered not suitable for FD using p64 MW HPC or p48 MW HPC.
* Aneurysm previously treated with a device in the parent vessel (e.g., stent, flow diverter).
* Another intracranial procedure scheduled for the following 6 months.
* Age < 18 years and > 80 years.
* Pregnancy possible or confirmed. Patient not able or willing to arrange contraception for 12 months after treatment.
* Patient not able or willing to adhere to the study protocol.
* Patient not able or willing to undergo the scheduled follow-up examinations.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The target population for this Observational Registry are patients with unruptured intracranial aneurysms suitable for flow diversion on operators' discretion. Patients can be included in the Observational Registry if they meet all of the inclusion and none of the exclusion criteria and have provided written informed consent.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2019-06-22 (Actual); Primary Completion 2023-06-22 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
Safety endpoint | Within 30 days after the intervention
  Occurence of ischemic or hemorrhagic stroke. Incidence of ischemic or hemorrhagic stroke in the territory supplied by the treated artery.

SECONDARY OUTCOMES:
Safety endpoint | Within the first 12 months after the intervention
  Occurence of all adverse events and serious adverse events, related directly or indirectly to the intervention, the used device or the required medication.

OTHER OUTCOMES:
Efficacy endpoint | 12 months after the intervention
  Complete occlusion or the neck remnant of the target aneurysm(s), identified by DSA (Digital subtraction angiography).

CONTACTS AND LOCATIONS:
Locations (1):
- Shastin Central Hospital, Ulaanbaatar, Bayangol District, Mongolia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Initial experience with the novel p64MW HPC flow diverter from a cohort study in unruptured anterior circulation aneurysms under dual antiplatelet medication — https://pubmed.ncbi.nlm.nih.gov/32640858/